CLINICAL TRIAL: NCT03537066
Title: Effect of Continuous Positive Airway Pressure Treatment for Obstructive Apnea on Phone Usage Habits: the Callsas Study
Brief Title: CALLSAS Study: Effect of Continuous Positive Airway Pressure Treatment for Obstructive Apnea on Phone Usage Habits
Acronym: CALLSAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inability to include subjects on schedule
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-A02540-53
Record Dates: First submitted 2018-03-28; First posted 2018-05-25 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPAP treatment (Other): All included OSA patients are going to be treated by CPAP
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — All patients included will be treated by CPAP

SUMMARY:
Continuous positive airway pressure (CPAP) treatment improves sleepiness, depression and social activities in patients with obstructive sleep apnea (OSA). This evolution can be captured from changes in phone usage habits coupled with a mobile-based services. The aim of this study is to assess the impact of CPAP treatment on phone usage habits in OSA patients.

DETAILED DESCRIPTION:
Callsas is a prospective study embarking newly diagnosed obstructive sleep apnea patients initiated to CPAP treatment.

The primary objective is to analyze the modifications in phone usage habits before and after CPAP treatment.

Secondary objectives:

* Correlation between changes in phone usage habits and evolution of sleepiness
* Correlation between changes in phone usage habits and evolution of depression scale
* Correlation between changes in phone usage habits and evolution of quality of life
* Correlation between changes in physical activity measured by phones and evolution of physical activity objectively measured by actigraphy and gait platform
* Correlation between phone usage habits and CPAP adherence

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed OSA patients initiated on CPAP
* Follow-up at home by AGIR à dom
* Customers of Orange (or Sosh) for mobile and/or fixed-line telephony for at least 6 months
* Patient who signed a written consent to participate in the study
* Patient affiliated to social security

Exclusion Criteria:

* Pregnant women
* Patients with disease not allowing to realize functional and locomotion tests
* Person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure (patient under guardianship or curatorship)
* Patient who, in the judgment of the investigator, may not be cooperative or respectful of the obligations inherent to participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Effect of CPAP on phone usage habits indices | from 6 months before CPAP treatment until 6 months after CPAP treatment initiation
  Changes in indices of phone usage habits

SECONDARY OUTCOMES:
Time course evolution of phone usage habits indices and evolution of sleepiness | from CPAP initiation until 6 months after CPAP treatment initiation
  Assessment of sleepiness by ESS
Time course evolution of phone usage habits indices and evolution of depression | from CPAP initiation until 6 months after CPAP treatment initiation
  Assessment of depression by Pichot scale
Time course evolution of phone usage habits indices and evolution of quality of life | from CPAP initiation until 6 months after CPAP treatment initiation
  Assessment of quality of life by SF-36
Time course evolution of phone usage habits indices and evolution of locomotion | from CPAP initiation until 6 months after CPAP treatment initiation
  patterns of locomotion objectively measured by a gait platform
CPAP adherence | from CPAP initiation until 6 months after CPAP treatment initiation
  Time course evolution of CPAP adherence assessed by telemonitoring versus time course evolution of phone usage habits
Access to care as a predictor of CPAP adherence | from CPAP initiation until 6 months after CPAP treatment initiation
  Care access questionnaire developed by ODENORE and National French insurance
Effect of food habit with CPAP treatment | At CPAP initiation and at 6 months after CPAP treatment initiation
  Changes in food frequence questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, Principal Investigator — CHU Grenoble Alpes
Locations (1):
- Grenoble Alps University Hospital, Grenoble, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: Undecided